CLINICAL TRIAL: NCT00360035
Title: A Multi-Center, Open-Label, Phase II Study of Single-Agent GX15-070MS Administered as a 24-Hour Infusion Every 2 Weeks to Patients With Myelofibrosis With Myeloid Metaplasia (MF)
Brief Title: Safety and Efficacy of Obatoclax Mesylate (GX15-070MS) in the Treatment of Myelofibrosis With Myeloid Metaplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM007
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GX15-070MS (Experimental): Obatoclax mesylate 60mg
  Interventions: Drug: Obatoclax mesylate (GX15-070MS)

INTERVENTIONS:
Drug: Obatoclax mesylate (GX15-070MS) — 60 mg q2wks

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogenic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase II study of single-agent obatoclax administered in 2-week cycles as a 24-hour infusion every 2 weeks at a fixed dose of 60 mg to patients with myelofibrosis. Infusions may be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described in the protocol may be administered with the intent to treat the patient's malignancy. Supportive care measures including those directed at controlling symptoms resulting from myelofibrosis (blood products, growth factor, hydroxyurea, etc.) are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed myelofibrosis with myeloid metaplasia.
* No limitations on allowable type and amount of prior therapy.
* Patients must have normal organ function.
* Must be willing to submit to blood sampling for planned PK and PD analyzes.
* Must have ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

* No other agents or therapies administered with the intent to treat malignancy.
* Patients with prior exposure to obatoclax.
* Uncontrolled, intercurrent illness.
* Pregnant women and women who are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2008-03 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determine the steady-state pharmacokinetic parameters and pharmacodynamic response. | 1 Year

SECONDARY OUTCOMES:
Peripheral blood counts | 4 Weeks to 1 Year
Bone marrow aspirates and biopsies | 8 weeks to 1 year
Transfusion and growth factor requirements | 8 weeks to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X, Inc.
Locations (7):
- United States (6):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Parikh SA, Kantarjian H, Schimmer A, Walsh W, Asatiani E, El-Shami K, Winton E, Verstovsek S. Phase II study of obatoclax mesylate (GX15-070), a small-molecule BCL-2 family antagonist, for patients with myelofibrosis. Clin Lymphoma Myeloma Leuk. 2010 Aug;10(4):285-9. doi: 10.3816/CLML.2010.n.059. PMID 20709666